CLINICAL TRIAL: NCT04552600
Title: A Randomized, Double-masked, Placebo-controlled Phase 1b/2a Study to Evaluate Clinical Efficacy and Safety of Nuvastatic™ in Patients With Non-proliferative Diabetic Retinopathy Without Center-involved Diabetic Macular Edema.
Brief Title: Study to Evaluate Clinical Efficacy and Safety of Nuvastatic™ - C5OSEW5050ESA in Diabetic Retinopathy.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Natureceuticals Sdn Bhd (Industry)
Collaborators: Ministry of Agriculture, Malaysia (Unknown); Quest International University, Malaysia. (Unknown); Advanced Medical and Dental Institute (AMDI), Universiti Sains Malaysia (Unknown); Universiti Sains Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIAG-CSP- 032
Record Dates: First submitted 2020-09-05; First posted 2020-09-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-masked, Placebo-controlled phase 1b/2a study
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NuvastaticTM 1000 mg (Experimental): NuvastaticTM 1000 mg(standardized extract of Orthosiphon Stamineus) will be given orally, three times per day for 12 months.
  Interventions: Drug: Nuvastatic
- Placebo (Active Comparator): NuvastaticTM (without active) will be given orally, three times per day for 12 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nuvastatic — Phase 1b Interventional, multi-centered, double-masked, randomized
  Other Names: Lanctos 75 standardized Orthosiphon Stamineus Extract
  Arms: NuvastaticTM 1000 mg
Other: Placebo — Phase 1b Interventional, multi-centered, double-masked, randomized
  Arms: Placebo

SUMMARY:
Diabetic retinopathy (DR) is a common complication of diabetes mellitus that leads to loss of vision and blindness among working age adults. An ideal adjunctive agent for treating DR hence should be polymorphic and possess antiangiogenic, neuroprotective, anti-inflammatory, anti-oxidant as well as anti-ischaemic properties.Natureceuticals Sdn Bhd assessed the efficacy of core ingredient of Nuvastatic™, Lanctos 75™ for the treatment and management of the diabetic retinopathic condition.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is a common complication of diabetes mellitus that leads to loss of vision and blindness among working age adults. During progression of DR, patients can develop diabetic macular edema (DME), which is characterized by the thickening of the macula caused by the breakdown of the blood-retinal barrier and consequent retinal vascular hyperpermeability. In 2010, the global prevalence of DR among adults with diabetes mellitus aged 20-79 years was estimated to be 34.6% for any DR and 6.81% for DME. DME is the leading cause of vision loss among patients with DR. It is associated with the type of diabetes, and increases with the duration and severity of disease. Other significant risk factors common to DR and DME include hyperglycemia and hypertension. DME negatively impacts patients' health-related quality of life and represents an economic burden due to the increased use of healthcare resources by affected patients.

In DR, which is a complex multifactorial disease, basically the retinal neovascularization occurs with the disturbance of physiological angiogenesis due to creation of hypoxic condition, which induces the oxygen demand in the retina (Roth, 1977; Smith et al., 1994; Chen and Smith, 2007). Consequently, in response to induced hypoxia, excessive production and over expression of VEGF and other pro-angiogenic factors take place in the retina. This ultimately induces the situation so called "pathological neovascularization" (Aiello et al., 1994; Folkman, 2006). Retinal ischemia is a common precursor to vitreal neovascularization in retinal diseases (Tolentino and Adamis, 1998) and is strongly associated with a local inflammatory response in the ischemic retina (Barouch et al., 2000).

While there is no curative treatment available for DME, laser photocoagulation represents an effective treatment to preserve vision. However, this treatment modality is limited by its inability to restore vision once it has been lost. The current standard of care for DME includes intravitreal anti-vascular endothelial growth factor (VEGF) therapeutics and corticosteroids. Clinical studies have confirmed that monthly intravitreal treatment with the anti-VEGF treatment can improve vision, with up to 45% of patients gaining ≥ 15 letters in best-corrected visual acuity (BCVA) after 24 months. Similar improvements were found after treatment with the anti-VEGF antibodies. Despite the proven efficacy of VEGF inhibitors, the requirement of frequent injections causes a high rate of treatment discontinuation among patients with DME and represents a major limitation.

Thus, current pharmacological treatments target single pathogenic processes with a narrow therapeutic range and may cause adverse side effects leading to undesired systemic effects. The presence of potential side effects and the significant proportion of patients who do not respond to treatment suggest that there remains a need for the development of improved therapies for DR and DME.

An ideal adjunctive agent for treating DR hence should be polymorphic and possess antiangiogenic, neuroprotective, anti-inflammatory, anti-oxidant as well as anti-ischaemic properties.

We have assessed the efficacy of core ingredient of Nuvastatic™, Lanctos 75™ for the treatment and management of the diabetic retinopathic condition. These scientific studies have shown that the standardized extract of O. stamineus (Lanctos 75™) in mediates antiangiogenic actions via blocking VEGF pathway. We demonstrated the potent antiangiogenic activity of the standardized extract of O. stamineus and prevention activity of the extract against human breast tumor in xenograft model. In addition, it is reported that, the extract was found to specifically inhibit VEGF expression and VEGFR phosphorylation known to be up-regulated in new blood vessel formation which in turn leads to suppression of vascularization and thereby ultimately the growth of tumor will be affected. Rosmarinic acid present in the extract could be involved in cell cycle arrest in the G0/G1 and G1/S phases, exhibiting an anti-proliferative effect of thus suggesting that the proliferative vascular diseases including retinopathy might be the potential target for the pharmacological application of rosmarinic acid. Also, the key active ingredients in the extract are rosmarinic acid mainly, and sinensetin, eupatorin and betulinic acid, which are readily absorbed into the plasma and exert that conferred the synergistic pharmacological response such as anti-inflammatory, antioxidant, analgesic and neuroprotective effects.

ELIGIBILITY:
Inclusion Criteria:

* • Type-2 Diabetes mellius (NIDDM) patients of both genders aged 18-65 years.

  * Able and willing to provide written informed consent.
  * Documented diagnosis of Type 2 diabetes mellitus a glycosylated hemoglobin A1c (HbA1c) of ≤ 12.0% at screening.
  * Patients preferably on oral medications for DM.
  * Meets specific ocular criteria for the study eye including but not limited to, the presence of non-proliferative diabetic retinopathy (NPDR) without center-involved diabetic macular edema (CI-DME) in the study eye at screening with NPDR level 47 or level 53, as determined by the central reading center (CRC) by using the DR severity scale (DRSS), for which treatment can be deferred for at least 4 weeks after Day 1 visit.
  * Media clarity, pupillary dilation, and subject cooperation sufficient to obtain adequate assessments. (Subject has early treatment diabetic retinopathy study (ETDRS) best corrected visual acuity (BCVA) letter score ≤ 73 (Snellen 20/40) and ≥ 24 (Snellen 20/320) at screening visit).
  * Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.

Study Eye Inclusion Criteria

* Best corrected E-ETDRS visual acuity letter score ≥74 (i.e.20/32 or better) within 8 days of randomization.
* On clinical exam, definite retinal thickening due to DME within 3000 μm of the center of the macula but not involving the central subfield.
* Thickened non-central macular subfields on spectral domain OCT macular map that meet either of the following criteria:

  1. At least two non-central macular subfields with OCT thickness above threshold (average normal + 2 SD) from DRCR.net approved spectral domain OCT machines- see below.
  2. At least one non-central macular subfield with OCT thickness at least 15 μm above threshold (average normal + 2 SD) from DRCR.net approved spectral domain OCT machines-see DRCR.net procedures manual for threshold details.
* Central subfield thickness <250 microns obtained by one of the following DRCR.net approved spectral domain OCT machines:

  1. Zeiss Cirrus
  2. Heidelberg Spectralis
  3. Optovue RTVue
* Media clarity, pupillary dilation, and study participant cooperation sufficient for adequate OCT and fundus photographs.
* If the study participant is on multiple ocular drops, investigator believes that study participant can be compliant with a multi-drop regimen.

Exclusion Criteria:

* Insulin dependent Diabetes mellitus (IDDM or T1DM) patients.
* Any condition that would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease or glycemic control).
* History of myocardial infarction or other acute cardiac event.
* History of chronic renal failure requiring dialysis or kidney transplant.
* Prior participation in any clinical study.
* Treatment with any investigational study drug within 30 days of screening.
* Known allergy to study product.
* Treatment with specific prohibited medications or therapy beginning 4 weeks prior to screening and throughout the duration of the study.
* Subject with macular edema considered to be due to a cause other than DME, decrease in BCVA due to causes other than DME, significant macular ischemia, any other ocular disease that may cause substantial reduction in BCVA, active peri-ocular or ocular infection.
* Subject with an history of following within 3 months prior to Day 1: non-infectious uveitis, high myopia (-8 diopter or more correction), pars plana vitrectomy, any ocular surgery, prior IVT, subtenon, or periocular, non-sustained release, steroid therapy, uncontrolled glaucoma,
* History of systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization.
* Any laboratory abnormalities at screening.
* Male subjects who are not surgically sterile and are not willing to practice a medically accepted method of birth control with their female partner of childbearing potential from screening through 30 days following completion of the study
* Female subjects of childbearing potential who are not willing to practice a medically accepted method of birth control with their non-surgically sterile male sexual partner from screening through 30 days following completion of the study
* Female subjects who are pregnant or lactating.
* Subject has media clarity, papillary constriction (i.e., senile miosis), or subject lacks cooperation that would interfere with any study procedures, evaluations or interpretation of data.
* Cataract surgery performed within 6 months prior to screening or planned during the trial; or any additional eye disease in the study eye that, in the opinion of the investigator, could compromise or alter visual acuity during the course of the study (e.g. vein occlusion, uncontrolled intraocular pressure (IOP) >24 mmHg on optimal medical treatment, glaucoma with visual field loss, uveitis or other ocular inflammatory disease, vitreomacular traction, monocular vision, history of ischemic optic neuropathy, or genetic disorders such as retinitis pigmentosa)
* Active center-involved DME (CI-DME) on clinical examination and Optical Coherence Tomography (OCT) central subfield thickness in the study eye above 300 μm as measured by Optovue OCT or above 320 μm as measured by Heidelberg OCT
* Anterior segment and vitreous abnormalities in the study eye that would compromise the adequate assessment of the best corrected visual acuity or an adequate examination of the posterior pole
* Evidence of neovascularization on clinical examination including active neovascularization of the iris (small iris tufts are not an exclusion) or angle neovascularization in the study eye, ruled out by gonioscopy (documented in the last 4 weeks before screening or performed at screening)
* Prior pan-retinal photocoagulation (defined as ≥ 100 burns placed previously outside of the posterior pole) in the study eye
* History of DME or DR treatment with macular laser within 3 months prior to screening, or intraocular injections of medication within 6 months prior to screening, and no more than 4 prior intraocular injections in the study eye at any time in the past
* Patients treated with Monoamine Oxidase (MAO) inhibitors or drugs that may have potential side effects due to MAO inhibition
* Current or planned, during the trial, use of medications known to be toxic to the retina, lens or optic nerve, or cause vision loss
* Patients who must or wish to continue the intake of other restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Estimated Glomerular filtration rate (eGFR) < 60 mL/min/1.73m2 calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at screening, or where the investigator expects filtration rate is likely to drop below 60 mL/min/1.73m2 during the trial
* Alanine transaminase (ALT) or aspartate transaminase (AST) greater than 2.0-fold the upper limit of normal, or total bilirubin > 1.5x upper limit of normal.
* Uncontrolled arterial hypertension defined as a single measurement of systolic blood pressure >180 mmHg, or two consecutive measurements of systolic blood pressure > 160 mmHg and/or diastolic blood pressure >100 mmHg on optimal medical regimen at screening. If blood pressure is brought to ≤ 160/100 mmHg by antihypertensive treatment until randomization, individual can become eligible.
* Wolff-Parkinson-White Syndrome, baseline QTc > 450 ms, family history of long QT, or on medication prolonging QT time at screening or planned initiation during the trial
* Diagnosis of a serious or unstable systemic or eye disease and other conditions that, in the clinical judgment of the investigator, are likely to interfere with the analyses of safety and efficacy in this study. Patients with an expected life expectancy of less than 2 years are also excluded.
* Active known or suspected chronic or relevant acute infections, such as HIV (Human Immunodeficiency Virus)\viral hepatitis, or tuberculosis. QuantiFERON® TB test and HBs Ag test will be performed during screening. Patients with a positive test result may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active infection.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable study participant or unlikely to complete the trial
* Known hypersensitivity to any component of the trial drug and/or allergy to fluorescein dye
* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomization or planned during the trial, e.g. hip replacement
* Currently enrolled in another investigational drug trial, or less than 30 days or 5 times half-life of the investigational drug, whichever is longer, since ending another investigational drug trial from the screening visit in this trial or receiving other investigational treatment(s); patients participating in a purely observational trial will not be excluded.
* Previous randomization in this trial
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Any other clinical condition that, in the opinion of the investigator, would jeopardize patient safety while participating in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy of Nuvastatic - Retinal Thickness | 12 months
  Central Subfield Retinal Thickness
To evaluate efficacy of Nuvastatic - protein biomarkers | 12 months
  protein biomarkers
To evaluate safety of Nuvastatic - Letter Score | 12 months
  Visual Acuity Letter Score

SECONDARY OUTCOMES:
To evaluate short-term visual outcomes on severity | 12 months
  effect of IP on severity of DR
To evaluate short-term visual outcomes on zone diagnosis | 12 months
  zone diagnosis
To evaluate short-term visual outcomes on DRSS | 12 months
  visual improvement DRSS

CONTACTS AND LOCATIONS:
Overall Officials: Aman Shah Abdul Majid, Ph.D., Principal Investigator — Quest International University
Locations (1):
- Fifepoint Multispeciality Hospital Pvt. Ltd., Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
Requested information by institutional researcher
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Completed study
Access Criteria: Institutional Researcher
URL: https://nature-ceuticals.com